CLINICAL TRIAL: NCT07273916
Title: Evaluation of the Efficacy and Onset of Action of a Topical Anesthetic Marker
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, Dr, Hexsel Dermatology Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-DPCHD-2025-05
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Pain Management
Keywords: anesthetic; analgesic; pain; control; topical
MeSH Terms: conditions — Agnosia; Pain | interventions — carbitol; Tetracaine; Lidocaine

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, self-controlled clinical study.
Masking Description: After cleansing the skin of the forearm selected by the participant (right or left), four points will be marked and the study product will be applied. Every 10 minutes, sensitivity at the application site and adjacent skin will be tested through superficial pricks performed with the same pressure in the treated area and the adjacent control area. The participant will be asked whether sensitivity is the same in both areas and will be requested to report the percentual reduction in pain at each studied point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention, self-controlled (Experimental): Self-controlled
  Interventions: Drug: Cutaneous marker (Transcutol P+ 20%, Tetracaine 7%, Lidocaine 23%, and dye q.s.),

INTERVENTIONS:
Drug: Cutaneous marker (Transcutol P+ 20%, Tetracaine 7%, Lidocaine 23%, and dye q.s.), — After cleansing the skin of the forearm selected by the participant (right or left), four points will be marked and the study product will be applied. Every 10 minutes, sensitivity at the application site and adjacent skin will be tested through superficial pricks performed with the same pressure in the treated area and the adjacent control area. The participant will be asked whether sensitivity is the same in both areas and will be requested to report the percentual reduction in pain at each studied point.

SUMMARY:
The goal of this clinical trial is to to demonstrate the efficacy of a topical anesthetic in reducing pain during the performance of a painful test on the participant's arm.

Primary Objective:

To evaluate the analgesic efficacy and onset of action of the cutaneous marker (Transcutol P+ 20%, Tetracaine 7%, Lidocaine 23%, and dye q.s.), assessed in comparison with a control area without anesthetic. Pain will be induced by light touches with the same pressure using a disposable needle tip on the forearm region, measured by a visual analog scale (VAS) at 10, 20, 30, and 40 minutes after application of the marker, in a sample of 20 participants.

● Secondary Objective: To assess safety through the recording

1. Methodology

   After cleansing the skin of the forearm selected by the participant (right or left), four points will be marked and the study product will be applied. Every 10 minutes, sensitivity at the application site and adjacent skin will be tested through superficial pricks performed with the same pressure in the treated area and the adjacent control area. The participant will be asked whether sensitivity is the same in both areas and will be requested to report the percentual reduction in pain at each studied point.
2. Proposed Evaluation Methods Visual Analog Scale (VAS).
3. Visits / Follow-up Duration The test will be conducted on the proposed area (forearm) during a single visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Willingness and ability to undergo the procedures described in the protocol.
3. Candidates who understand and sign the Informed Consent Form (ICF) upon study entry, prior to any study-related procedures.

Exclusion Criteria:

1. Pregnant or breastfeeding on the day of the study.
2. History of sensitivity to topical anesthetics or any component of the anesthetic marker formulation.
3. Symptoms of infection at the application site.
4. Eczema or skin alterations at the application site.
5. Any other active inflammations or infections in the treated areas.
6. Any surgical procedure performed that may have affected the area to be assessed in this study.
7. Severe psychiatric disorders.
8. Any other uncontrolled chronic or serious medical condition which, in the investigator's opinion, may interfere with the interpretation of the clinical study results or place the participant at significant risk.
9. Use of analgesic medications.
10. Vulnerable groups (such as individuals deprived of liberty) as defined in Section 1.61 of the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines.
11. Participation in any other clinical drug or device study and/or participation within 7 days prior to Day 1 of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain control | 1 day
  To evaluate, record, and compare mean Visual Analog Scale (VAS) scores at 10-minute intervals, with time 0 corresponding to product application and the first assessment occurring 10 minutes after application, followed by measurements at 20, 30, and 40 minutes.
  Assessments will be performed on the left or right forearm according to the participant's preference, using light punctures in the area where the product was applied and comparing results to an adjacent control area.

SECONDARY OUTCOMES:
Time to analgesic effect | 1 day
  Onset of analgesic effect, defined as the first clinically relevant reduction in VAS pain scores following product application.
  ● Difference in pain scores between puncture points in the untreated control area and the treated area, assessed at the same time points.